CLINICAL TRIAL: NCT06022731
Title: A Yolo-V5 Approaches to Evaluation of Filling and Overhanging Filling: An Artificial Intelligence Study
Brief Title: Artificial Intelligence Evaluation of Fillings
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Elif Bilgir, Associated Professor, Eskisehir Osmangazi University
Other Study IDs: Retrospective
Record Dates: First submitted 2023-08-08; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Dentomaxillofacial Radiology
Keywords: dental filling; dentistry; deep learning,
MeSH Terms: interventions — Radiography, Panoramic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Filling
  Interventions: Diagnostic Test: Panoramic Radiography
- Overhanging Filling
  Interventions: Diagnostic Test: Panoramic Radiography

INTERVENTIONS:
Diagnostic Test: Panoramic Radiography — this retrospective study includes analysis of radiographs previously taken from patients for various purposes

SUMMARY:
The goal of this Non-Interventional Clinical Research is to detect the prevalence and distribution of filling and overhanging filling without the need for additional bitewing radiographs using panoramic images, based on a deep CNN (Convolutional Neural Network) architecture trained through supervised learning.

In this study, retrospectively obtained radiographs were used in the development of artificial intelligence models for relevant situations. These datasets were obtained from the images of the patients who applied to ESOGU (Eskişehir Osmangazi University) Dentistry Faculty, Dentomaxillofacial Radiology clinic for various dental purposes. Eskisehir Osmangazi University Non-Interventional Clinical Research Ethics Board (decision date and decision number: 04.10.2022/22) approved the study protocol. The principles of the Helsinki Declaration were followed in the study.

ELIGIBILITY:
Inclusion Criteria:

* Images of individuals in the permanent dentition period
* Artifact-free images in the examination region
* Individuals with a history of restorative dental treatment

Exclusion Criteria:

* Images of individuals in mixed dentition
* Radiographic images obtained by incorrect positioning of the patient or containing artifacts

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: These datasets were obtained from the images of the patients who applied to ESOGU Dentistry Faculty, Dentomaxillofacial Radiology clinic for various dental purposes.
Sampling Method: Probability Sample
Enrollment: 4323 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
The success of artificial intelligence models for filling and overhanging filling | 1 year
  It is obtained by calculating the sensitivity, precision, and F1 scores values for filling and overhanging filling.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskişehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to publish the findings obtained as a result of the study in internationally journals and share this information within the publication.
Supporting Information: Study Protocol, SAP, CSR